CLINICAL TRIAL: NCT03013673
Title: Predicting Visceral Leishmaniasis in HIV Infected Patients
Acronym: PreLeisH
Status: Terminated | Type: Observational
Why Stopped: Due to the ongoing conflict in the Tigray region
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University of Gondar, Gondar, Ethiopia (Unknown); Medecins Sans Frontieres, Netherlands (Other); Bureau of Health, Abdurafi, Ethiopia (Unknown)
Responsible Party: Sponsor
Other Study IDs: ITM0915
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Leishmaniasis, Visceral
Keywords: leishmaniasis, visceral, neglected, HIV, co-infection, asymptomatic, Ethiopia
MeSH Terms: conditions — Leishmaniasis, Visceral; Leishmaniasis; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All samples and sample left-overs (blood and urine) not used during the course of this study will be stored for 25 years after the end of the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV: HIV infected individuals residing in VL-endemic areas in Northern Ethiopia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In this cohort study, the investigators will study the asymptomatic period preceding the onset of active Visceral Leishmaniasis (VL) in HIV-infected individuals from VL endemic regions in Ethiopia as an avenue to develop an evidence-based screen and treat strategy to prevent progression to active VL.

DETAILED DESCRIPTION:
HIV co-infection drastically increases the risk of developing active VL. Clinical outcomes are dire in immune-compromised patients even with the best available treatment, and relapse is frequent. The incubation period may provide an important window of opportunity for a pre-emptive "screen an treat" approach in HIV co-infected patients to prevent progression from infection to the active disease. However, no recommendations exist to date due to lack of solid evidence.

It is not known which patients are at highest risk of disease progression, which role parasite/host/HIV factors play in the asymptomatic infection phase, and what the diagnostic values of existing Leishmania infection markers are. Such information is needed to develop a prognostic clinical tool for the detection of HIV patients at high risk of developing active VL.

Therefore, the aim is to study the asymptomatic period preceding the onset of active VL in HIV-infected individuals from VL endemic regions in Ethiopia as an avenue to develop an evidence-based screen and treat strategy to prevent progression to active VL. This will be a prospective cohort study with one year of follow-up for patients who remain VL free. Patients developing active VL during the study period will be followed until the end of the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-positive
* Enrolled in HIV care at the study site

Exclusion Criteria:

* Age under 18 years
* Diagnosis of active Visceral Leishmaniasis at enrolment
* Unlikely to seek health care again at this site during the next two years
* Not able or willing to provide informed consent. For patients not able to provide informed consent: No guardian available or willing to provide IC
* Medical emergency, underlying chronic medical condition, or other circumstances that make adherence to the study unlikely, or participation in the study medically inadvisable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals residing in VL-endemic areas in Northern Ethiopia
Sampling Method: Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of asymptomatic Leishmania infection | January 2018
  The proportion of individuals with asymptomatic Leishmania infection at enrolment, among all enrolled participants
Incidence rate of asymptomatic Leishmania infection | January 2020
  The number of individuals with newly diagnosed asymptomatic Leishmania infection per person-years at risk during follow-up, among participants without Leishmania infection at enrolment
Evolution of Leishmania infection markers | January 2020
  The proportions of individuals with positive test results for the different Leishmania infection markers at each follow-up visit
Incidence rate of active VL | January 2020
  The number of individuals who develop active VL per person-years at risk during follow-up, among all enrolled participants
Risk factors for active VL | January 2020
  The association between the risk to develop active VL during follow-up and demographic/clinical characteristics as well as HIV/host immunity/Leishmania infection markers from baseline onwards
Prognostic tool for active VL | January 2021
  A clinical decision algorithm, prioritizing and integrating identified risk factors, that is able to most efficiently predict the risk of developing active VL within 12 months

SECONDARY OUTCOMES:
Patterns in host immune markers for asymptomatic Leishmania infection | January 2020
  The association between asymptomatic Leishmania infection and the levels of the different host immune markers, among participants tested for host immune markers
Evolution of host immune markers | January 2020
  The average levels of the different host immune markers at each follow-up visit
Patterns in host immune markers for VL treatment failure | January 2021
  The association between the risk of VL treatment failure and the levels and evolution of the different host immune markers, among participants who develop active VL and receive VL treatment
Patterns in host immune markers for VL relapse | January 2021
  The association between the risk of VL relapse and the levels and evolution of the different host immune markers, among participants who develop active VL

CONTACTS AND LOCATIONS:
Overall Officials: Johan van Griensven, MD PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium; Ermias Diro, MD, Study Director — College of Medicine and Health Sciences, University of Gondar, Gondar, Ethiopia
Locations (1):
- Abdurafi Health Center, Ābderafī, Amhara, Ethiopia